CLINICAL TRIAL: NCT01183364
Title: A Phase 1, Pharmacokinetic Study of STA-9090 in Combination With Docetaxel in Subjects With Advanced Solid Tumor Malignancies
Brief Title: A Dose Escalation Study of STA-9090 and Docetaxel in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9090-07
Record Dates: First submitted 2010-08-11; First posted 2010-08-17 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Solid Tumor Malignancies
Keywords: solid tumor malignancies; tumor; cancer; STA-9090; ganetespib; HSP90 inhibitor
MeSH Terms: conditions — Neoplasms | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STA-9090 and Docetaxel (Experimental): STA-9090 (ganetespib) and Docetaxel
  Interventions: Drug: STA-9090 (ganetespib) with Docetaxel

INTERVENTIONS:
Drug: STA-9090 (ganetespib) with Docetaxel — One treatment cycle will consist of weekly treatments for 2 weeks followed by a 1-week rest period. Treatment cycles will be repeated every 3 weeks. STA-9090 will be administered on Days 1 and 8 of each cycle and docetaxel will be administered on Day 1 of each cycle. Each agent will be administered as a separate 1-hour intravenous infusion.

SUMMARY:
This is an open-label, Phase 1, dose-escalation study to determine the recommended doses of STA-9090 (ganetespib) and docetaxel for the treatment of subjects with solid tumor malignancies. The safety and tolerability of the treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed metastatic or unresectable malignancy with evidence of progression
* If subject has been treated with docetaxel, must have evidence of persistent or progressive disease
* Measurable disease per RECIST
* CNS metastases are permitted if treated and radiographically and clinically stable for 4 weeks prior to first dose
* ECOG status less than or equal to 2
* Life expectancy greater than 3 months
* Adequate hematological, hepatic and renal function as defined by protocol
* Willingness and ability to comply with study requirements
* Female subjects of childbearing age must have a negative pregnancy test at study entry
* Female subjects of child bearing age and males must agree to use adequate contraception as defined in the protocol

Exclusion Criteria:

* Prior chemotherapy or investigational agents within 3 weeks or 5 times the agent's half life, whichever is shorter prior to first dose
* Radiotherapy within 2 weeks of first dose
* Surgery, radiotherapy or ablative procedure to the only area of measurable disease
* Major surgery within 4 weeks of first dose
* Poor venous access that would require an indwelling catheter for study drug administration
* History of severe allergic or hypersensitivity reactions to STA-9090 or docetaxel or their diluents or excipients
* Baseline QTc >470 msec or previous history of QT prolongation while taking other medications
* Peripheral neuropathy > Grade 1
* Ventricular ejection fraction less than or equal to 55% at baseline
* Treatment with chronic immunosuppressants. However subjects may receive steroids for stable CNS metastases
* Women who are pregnant or lactating
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety of STA-9090 (ganetespib) and docetaxel combination | June 2011
  The number of adverse events will be used as a measure of safety

SECONDARY OUTCOMES:
Pharmacokinetics | June 2011
  Pharmacokinetics of STA-9090 (ganetespib) and Docetaxel. This includes concentrations of these drugs in patients' blood at various protocol-specified times relative to the time of dose administration. These will be summarized by parameters including maximum concentration, total exposure and how fast the patient's body gets rid of the drug (known as Cmax, AUC, t1/2, respectively).

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States